CLINICAL TRIAL: NCT05811728
Title: Three-dimensional Assessment of the Bone Changes Accompanying Laser-assisted Orthodontic Tooth Movement: a Randomized Controlled Clinical Trial
Brief Title: Three-dimensional Assessment of the Bone Changes Accompanying Laser-assisted Orthodontic Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: #202
Record Dates: First submitted 2023-04-01; First posted 2023-04-13 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Low Level Laser Therapy; Canine Retraction; Orthodontic Tooth Movement
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled clinical trial, involving the split-mouth design, with one side of the maxillary arch serving as the control group, and the other side serving as the experimental group.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low level laser therapy (Experimental)
  Interventions: Radiation: Low level laser therapy
- Control (Placebo Comparator)
  Interventions: Other: without beam emission

INTERVENTIONS:
Radiation: Low level laser therapy — The low-level laser applied will be a Diode laser* emitting infrared radiation at a wavelength of 980 nm, in a continuous mode. On the experimental side, subjects will receive LLLT on days 0, 3, 7, 14, and every 2 weeks thereafter, till the termination of the study period (3 months).
  Arms: Low level laser therapy
Other: without beam emission — The laser tip will be held passively on the control side without beam emission, providing a placebo effect.
  Arms: Control

SUMMARY:
Aim of the present study is to evaluate the effect of low-level laser therapy on bone quality and quantity with orthodontic tooth movement.

ELIGIBILITY:
Inclusion Criteria:

* Malocclusion that requires at least the extraction of maxillary first premolars, followed by canine retraction into the extraction site, such as Class I bimaxillary protrusion, and Class II division 1 cases.
* Normal shape and structure of the maxillary canines, with no history of root canal treatment

Exclusion Criteria:

* Patients who underwent previous orthodontic treatment.
* Patients currently receiving drug therapy, e.g. hormonal therapy and corticosteroids, as well as patients with chronic diseases.
* Pregnancy and lactation.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-25 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Measurement of alveolar bone density | 3 months
  Bone density will be measured from cone beam computed tomography (CBCT) scans at 2 different locations on each side of the upper arch; between the canine and lateral incisor, and between the canine and second premolar. Bone density will be measured using Hounsfield Units (HU).
Measurement of alveolar bone microstructure | 3 months
  From the CBCT scans, the maxillary alveolar process between the canine and lateral incisor, and between the canine and second premolar will be examined. Bone microstructures will be measured and calculated with a dedicated software.
Measurement of buccal bone thickness | 3 months
  buccal bone thickness will be measured from the CBCT scans. Three points will be measured from the buccal bone to the root, at the coronal, mid-root, and apical level
Measurement of alveolar bone volume | 3 months
  From CBCT scans, bone volume in areas of the maxillary alveolar process between the canine and lateral incisor, and between the canine and second premolar will be measured
Measurement of bone Microstructure | 3 months
  Using the collected CBCT scans, the region of interest will be selected within the maxillary alveolar process, and fractal dimension analysis will be performed using a special software.

CONTACTS AND LOCATIONS:
Overall Officials: Farah Y Eid, PhD, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt